CLINICAL TRIAL: NCT01659125
Title: Effectiveness and Neuropsychological Predictors of Guided Self-Help for OCD
Brief Title: Effectiveness and Neuropsychological Predictors of Guided Self-Help for Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIEF003581HI
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OCFighter (Experimental): OCFighter
  Interventions: Behavioral: "OCFighter"

INTERVENTIONS:
Behavioral: "OCFighter" — OCFighter™ s an interactive, internet guided self-help (GSH) treatment program for obsessive-compulsive disorder (OCD). It uses the evidence based approach known as Cognitive Behavioral Therapy (CBT) and was adapted from the previously validated BT STEPS program for OCD. The program teaches the best practice CBT technique to help with OCD called exposure with ritual prevention (ERP).
  Other Names: OCFighter; Guided Self-help

SUMMARY:
The primary aim of this study is to learn about who is most likely to benefit from guided self-help (GSH) for obsessive-compulsive disorder (OCD).

DETAILED DESCRIPTION:
40 Participants with OCD will be recruited. They will be given access to OC Fighter, an internet OCD treatment program. During the 17 week program, participants will meet with a therapist 9 times. Assessments will occur at pretreatment, post-treatment, 3-month follow up and 6-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Principal or co-principal diagnosis of OCD
* Clinical global impression score greater than or equal to 4
* Y-BOCS score great than or equal to 8
* Fluency in English
* Capacity to understand the nature of the study and willingness to sign informed consent form

Exclusion Criteria:

* Active manic episode, psychosis, pervasive developmental disorder, mental retardation
* Concurrent OCD psychotherapy
* Current threat of harm to self or others
* Previous adequate trial of therapist-administered or self-administered exposure and response prevention for OCD

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Diefenbach, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- OCFighter Participants: OCFighter
  "OCFighter": OCFighter™ s an interactive, internet guided self-help (GSH) treatment program for obsessive-compulsive disorder (OCD). It uses the evidence based approach known as Cognitive Behavioral Therapy (CBT) and was adapted from the previously validated BT STEPS program for OCD. The program teaches the best practice CBT technique to help with OCD called exposure with ritual prevention (ERP).
Period: Overall Study
Arm/Group | OCFighter Participants
Started | 26
Initiated Treatment | 24
Completed the Posttreatment Assessment | 17
Completed 3-month Follow-up | 16
Completed 6-month Follow-up | 12
Completed | 12
Not Completed | 14
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 7
Not completed — Technical Problem | 1
Not completed — Time Constraints | 2
Not completed — Failed to Start Treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | OCFighter Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.08 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)
Description: The Y-BOCS is a semi-structured interview that assesses severity of obsessions and compulsions. The total score is reported here and ranges from 0 to 40 with higher scores indicating more severe OCD symptoms.
Time Frame: Baseline (pretreatment), 17-weeks (posttreatment), and 6 month-follow-up
Population: Results are reported at each time-point for the intent-to-treat sample of participants who initiated treatment (n = 24).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OCFighter Participants: Participants who initiated treatment
Arm/Group | OCFighter Participants
Number analyzed (Participants) | 24
units on a scale
  Baseline (pre-treatment) | 24.67 (5.16)
  week 17 (post-treatment) | 18.29 (9.06)
  6-month Follow-up | 18.46 (7.79)

2. Primary Outcome: Responder Status
Description: Participants who experienced a clinically significant change in Y-BOCS score defined as posttreatment YBOCS score that (a) has decreased by a reliable level (at least 1.96 times the standard deviation of that measure, taking into account the reliability of the measure itself; in this case, a decrease of 5 points or more), and (b) is within the nonclinical range of scores (in this case, a score of 13 or below).
Time Frame: Week 17 (post-treatment) and 6-month follow-up
Population: Results are reported at each time-point for the intent-to-treat sample of participants who initiated treatment (n = 24).
Measure: Number; unit: participants
Arm/Group | OCFighter Participants
Number analyzed (Participants) | 24
participants
  Week 17 (post-treatment) | 5
  6- Month follow-up | 5

ADVERSE EVENTS:
Arm/Group | OCFighter Participants
Serious Adverse Events (participants affected / at risk) | 1/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCFighter Participants (N=24)
Increased Depression (Psychiatric disorders) | 1 (1) — There was one serious adverse event with a patient hospitalized for increased depression and suicidal ideation following onset of an acute psychosocial stressor which was unrelated to OCD symptoms

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No